CLINICAL TRIAL: NCT06125002
Title: Evaluation of the Prophylactic Effects of the Flavonoid Diosmin on Delayed-onset Muscle Soreness in Humans: a Randomized, Double-blinded and Placebo-controlled Single-center Clinical Trial
Brief Title: Diosmin for Treatment of Delayed-onset Muscle Soreness (DOMS)
Acronym: UEL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sergio Marques Borghi (Other)
Collaborators: Universidade Norte do Paraná (Other)
Responsible Party: Sponsor-Investigator, Sergio Marques Borghi, Principal investigator, Universidade Estadual de Londrina
Organization: Universidade Estadual de Londrina (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 64025122.2.0000.0108
Record Dates: First submitted 2023-10-20; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Myalgia
Keywords: delayed-onset muscle soreness; DOMS; exercise; flavonoids; diosmin
MeSH Terms: conditions — Myalgia; Motor Activity | interventions — Diosmin; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (placebo, corn starch tablets) (Experimental): Treatment will occur by oral route, and everyone will ingest identical opaque capsules (750 mg). The treatment protocol will be applied before the start (pre-treatment) of the intense dynamic exercise sessions, once a day, during the two days before, and on the day (immediately before) the execution of the exercise protocol.
  Interventions: Drug: Placebo
- Intervention (diosmin) (Experimental): Treatment will occur by oral route, and everyone will ingest identical opaque capsules (750 mg). The treatment protocol will be applied before the start (pre-treatment) of the intense dynamic exercise sessions, once a day, during the two days before, and on the day (immediately before) the execution of the exercise protocol.
  Interventions: Drug: Diosmin750

INTERVENTIONS:
Drug: Diosmin750 — The ingestion will occur orally, under monitoring by the responsible investigator.
  Other Names: Diosmine
  Arms: Intervention (diosmin)
Drug: Placebo — The ingestion will occur orally, under monitoring by the responsible investigator.
  Other Names: Corn starch tablets
  Arms: Intervention (placebo, corn starch tablets)

SUMMARY:
The potential benefits of exercise for the treatment of chronic inflammatory diseases and pain have been well documented in the scientific literature. Psychiatric, neurological, metabolic and cardiovascular diseases are examples of conditions that impact the health and quality of life of the population. Due to the effects provided by exercise, it can modify the natural course of these diseases. This concept is important to justify the efforts made by government bodies committed to promoting exercise, such as the WHO. However, the habitual practice of physical activity following the primary guidelines may be hampered by some factors, including those that support the physiological repercussions of exercise on the body, such as muscle pain. In this sense, an important complicating factor such as delayed-onset muscle soreness (DOMS), present in the post-exercise recovery period, can impair adherence and permanence in physical activity programs, thus representing a considerable barrier to exercise promotion. They can also severely impair the performance of high-level athletes. Flavonoids, present in plants, but also in foods of the human diet, are known to have several biological properties, including analgesic, anti-inflammatory, and antioxidant effects. Currently, there are still few studies that have evaluated the effects of flavonoids on the development and evolution of DOMS in humans.

DETAILED DESCRIPTION:
Main objective:

• Analyze the potential effects of supplementation with the flavonoid diosmin on DOMS in humans (athletes from the women's five-a-side soccer team from the city of Londrina, Paraná State, Brazil), using the proposed intense dynamic exercise protocol.

Specific objectives:

* Evaluate whether treatment with the flavonoid diosmin reduces muscle pain induced by the intense dynamic exercise protocol;
* Evaluate whether treatment with the flavonoid diosmin reduces systemic (serum) levels of total creatine phosphokinase (CFQ) and oxidative stress (lipid peroxidation and antioxidant capacity) induced by the intense dynamic exercise protocol;
* Evaluate whether treatment with the flavonoid diosmin is capable of improving the reduction in muscular performance and impairment of balance induced by the intense dynamic exercise protocol.

The present project will be carried out through a randomized, double-blinded and placebo-controlled clinical study. A total of approximately 40 female athletes pertaining to the Londrina Esporte Clube (name in Portuguese of the team) women's five-a-side soccer will be recruited for the study. The choice of exclusively women individuals is due to sexual dimorphism in pain perception, thus contributing to the results being more homogeneous and reliable. The criteria for inclusion of volunteer participants in the project will be to be between 16 and 35 years old, and to be able to perform the proposed intense dynamic exercise protocol. Exclusion criteria will include locomotor system dysfunctions or use of analgesic/anti-inflammatory medication at the time of recruitment, as well as being on a calorie-restricted diet or ergogenic supplementation. The study will consist of two experimental groups, made up of healthy individuals, who will perform the proposed intense dynamic exercise protocol, as follows: 1) control group that will receive placebo supplementation (corn starch tablets at a concentration of 750 mg); and 2) intervention group that will receive supplementation with diosmin (tablets at a concentration of 750 mg). Treatment of study participants will occur orally, and everyone will ingest identical opaque capsules containing placebo or diosmin with water. The treatment protocol will be applied before the start (pre-treatment) of the intense dynamic exercise sessions, once a day, during the two days before, and on the day (immediately before) the execution of the exercise protocol. Each experimental group will consist of approximately 20 participants. The project is approved by the Research Ethics Committee (CEP) for Human Beings/Brazil Platform(protocol number 64025122.2.0000.0108). The selected participants will be informed about the objectives and methodology of the study and when there is agreement with the proposed design, the agreement to voluntarily participate in the study will be registered by means of an Informed Consent Form. The intense dynamic exercise modality proposed (concentric and eccentric contractions) for the study will follow the following approach: participants will perform a standardized muscle injury protocol that will consist of a sequence of three sets of repetitions until fatigue of bilateral muscle contractions on a leg-press machine with a 45° angle. Each The participant will have their load previously defined through the 1 repetition maximum (1RM) test, and 70% of the defined weight will be used during the intense dynamic exercise protocol. During each action, the load will be resisted with the legs placed on the leg-press supporter from full knee extension to the 90° knee flexion angle, lasting approximately 3-5 seconds. Between each series, participants will be able to take a 1-minute rest period. The intense dynamic exercise protocol that will be carried out by all participants will be supervised by the project manager and/or collaborators duly trained for such assessments. Participants' clinical signs will be monitored frequently during the activities and in case of discomfort, the activity will be stopped immediately. Analyzes of clinical and blood parameters will be carried out before the start (baseline) and after the end of the proposed intense dynamic exercise protocol (24 and 48 hours) aiming to investigate the possible effects of diosmin on DOMS and related pathological events.

ELIGIBILITY:
Inclusion Criteria:

* Be within the pre-determined age range.
* Be able to perform the proposed intense dynamic exercise protocol.

Exclusion Criteria:

* Locomotor system dysfunctions.
* Use of analgesic/anti-inflammatory medication at the time of recruitment.
* Calorie-restricted diet or ergogenic supplementation.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Muscle soreness | Basal, 24, and 48 hours after DOMS induction protocol
  Evaluated by both digital algometer (in kilograms force; Kgf) and visual analogue (VAS) scale (in centimeters; cm), where 0 represents no pain and 10 the worst possible pain.

SECONDARY OUTCOMES:
Muscle tissue damage through the evaluation of the creatine phosphokinase (CPK) levels. | Basal, 24, and 48 hours after DOMS induction protocol
  Evaluated by spectrophotometric analysis using commercial kits (in milligram per liter; mg/L)
Plasmatic lipid peroxidation levels | Basal, 24, and 48 hours after DOMS induction protocol
  Evaluated by spectrophotometric analysis (in micromol per liter; µmol/L).
Plasmatic total antioxidant status | Basal, 24, and 48 hours after DOMS induction protocol
  Evaluated by spectrophotometric analysis (in millimol per liter; mmol/L).
Recovery of muscle function through the evaluation of the average and maximum torque of the knee extension for determining quadriceps strength (maximum voluntary isometric contraction; MVIC). | Basal, 24, and 48 hours after DOMS induction protocol
  Evaluated by isometric dynamometer (flexor/extension chair, in newton per meter; N/m).
Recovery of muscle function through vertical jump height. | Basal, 24, and 48 hours after DOMS induction protocol.
  Evaluated by jump strength (in milliseconds; msec).
Bipedal and single-legged (unipedal) postural balance. | Basal, 24, and 48 hours after DOMS induction protocol.
  Evaluated through the antero-posterior (AP) and mediolateral (ML) displacement velocities (in centimeter per seconds; cm/sec).

CONTACTS AND LOCATIONS:
Overall Officials: Sergio M Borghi, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luque MZ, Aguiar AF, da Silva-Araujo AK, Zaninelli TH, Heintz OK, Saraiva-Santos T, Bertozzi MM, Souza NA, Junior EO, Verri WA Jr, Borghi SM. Evaluation of a preemptive intervention regimen with hesperidin methyl chalcone in delayed-onset muscle soreness in young adults: a randomized, double-blinded, and placebo-controlled trial study. Eur J Appl Physiol. 2023 Sep;123(9):1949-1964. doi: 10.1007/s00421-023-05207-2. Epub 2023 Apr 29. PMID 37119360
- [Background] Borghi SM, Zaninelli TH, Saraiva-Santos T, Bertozzi MM, Cardoso RDR, Carvalho TT, Ferraz CR, Camilios-Neto D, Cunha FQ, Cunha TM, Pinho-Ribeiro FA, Casagrande R, Verri WA Jr. Brief research report: Repurposing pentoxifylline to treat intense acute swimming-Induced delayed-onset muscle soreness in mice: Targeting peripheral and spinal cord nociceptive mechanisms. Front Pharmacol. 2023 Jan 10;13:950314. doi: 10.3389/fphar.2022.950314. eCollection 2022. PMID 36703752
- [Background] Bussulo SKD, Ferraz CR, Carvalho TT, Verri WA Jr, Borghi SM. Redox interactions of immune cells and muscle in the regulation of exercise-induced pain and analgesia: implications on the modulation of muscle nociceptor sensory neurons. Free Radic Res. 2021 Jul;55(7):757-775. doi: 10.1080/10715762.2021.1953696. Epub 2021 Jul 19. PMID 34238089
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Heiss R, Lutter C, Freiwald J, Hoppe MW, Grim C, Poettgen K, Forst R, Bloch W, Huttel M, Hotfiel T. Advances in Delayed-Onset Muscle Soreness (DOMS) - Part II: Treatment and Prevention. Sportverletz Sportschaden. 2019 Mar;33(1):21-29. doi: 10.1055/a-0810-3516. Epub 2019 Mar 13. PMID 30865998
- [Derived] da Cunha FCB, Cortez GB, Pucci IM, Silva MM, Borim JM, Bertozzi MM, Jacinto JL, Carvalho TT, Aguiar AF, Casonatto J, Junior EO, Verri WA Jr, Borghi SM. Effects of the Flavonoid Diosmin on Post Exercise Muscle Soreness - A Randomized Controlled Trial. J Diet Suppl. 2025;22(6):977-998. doi: 10.1080/19390211.2025.2547167. Epub 2025 Aug 16. PMID 40818103